CLINICAL TRIAL: NCT00970515
Title: A Prospective, Multicenter, Randomized Trial Comparing Laparoscopy VS Conventional Mesh Repair of Incisional and Umbilical Hernia
Brief Title: Laparoscopic or Conventional Mesh Repair of Incisional and Umbilical Hernia
Acronym: EVENTRALAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recrutment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K060214; 2007-A00374-49 (Other: IDRCB)
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Incisional Hernia; Umbilical Hernia
Keywords: Laparoscopy; Incisional hernia; Umbilical hernia; Mesh repair; Postoperative complications
MeSH Terms: conditions — Incisional Hernia; Hernia, Umbilical; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic approach (Experimental): group A: Laparoscopic approach
  Interventions: Procedure: Laparoscopic mesh hernia repair
- Open approach (Active Comparator): group B: Open anterior approach
  Interventions: Procedure: Open anterior approach

INTERVENTIONS:
Procedure: Laparoscopic mesh hernia repair — The mesh is intraperitoneal
  Other Names: laparoscpic mesh repair of incisional and umbilical hernia
  Arms: Laparoscopic approach
Procedure: Open anterior approach — The mesh is placed by an anterior approach. It is placed after incision of the skin over or under the abdominal muscles, or is intraperitoneal
  Other Names: Conventional treatment of incisional and umbilical hernia
  Arms: Open approach

SUMMARY:
The aim of this study is to compare immediate and long-term (24 months) results of laparoscopic and open mesh repair of incisional and umbilical hernia.

DETAILED DESCRIPTION:
The aim of this study is to compare immediate and long-term (24 months) results of laparoscopic and open mesh repair of incisional and umbilical hernia.

Five hundred patients will be included in this randomized, multicentric trial.

Hypotheses are that laparoscopic approach: 1- reduces immediate parietal complications without increasing intra abdominal septic complications 2- is less invasive and also reduces patients' hospital stay and recovery time; 3- has the same efficacy, than open approach.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Incisional or umbilical hernia over 2 cm and less than 6 cm in diameter

Exclusion Criteria:

* Patients with a complicated incisional (pain, occlusion, cutaneous necrosis), irreductible painless incisional or umbilical hernia will not be considered as a complication
* Patients with a recurrence of incisional hernia
* Patients with an incisional or umbilical hernia whose lateral edges are located so that fixation of the mesh (which must extend beyond the 4 to 5 cm) is not possible
* Pregnant women
* Patients with HIV therapy
* Patients with cirrhotic ascites or other signs of hepatic insufficiency (bilirubin> 35 micromol / l; TP < 55%) or significant thrombocytopenia (< 60 000 platelets)
* Patients with a contra indication for laparoscopy
* Patients with a life expectancy < one year, or whose mobility within two years of treatment will damage proper monitoring
* Patients unable to understand information about the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Parietal postoperative complications: 1- haematoma, 2- abscess, 3- seroma 4- cutaneous necrosis | 2 months
Postoperative intra abdominal complications: peritonitis, occlusion, haemorrhage | 2 months

SECONDARY OUTCOMES:
Postoperative pain: measured by a- Visual Analogic Score (VAS 0-10): 1-number of days with VAS > 5; 2- maximal VAS, and b- duration (days) of morphine use | 2 months
Postoperative fever > 38°5 | 2 months
Postoperative ileus | 2 months
Postoperative phlebitis | 2 months
Postoperative pulmonary embolism | 2 months
Postoperative urinary infection | 2 months
Duration of hospital stay | 2 months
Duration of drainage | 2 months
Mesh infection | 24 months
Peritonitis due to intraperitoneal mesh | 24 months
Occlusion due to intra peritoneal mesh | 2 months
Recurrence of incisional or umbilical hernia | 24 months
Trocar site hernia | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Ms Vons, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Jean Verdier, department of digestive and general surgery, Bondy, France

REFERENCES:
- [Background] Slim K, Vons C. [Inguinal hernia repair: results of randomized clinical trials and meta-analyses]. J Chir (Paris). 2008 Mar-Apr;145(2):122-5. doi: 10.1016/s0021-7697(08)73720-7. French. PMID 18645551
- [Background] Vons C. [Laparoscopic treatment of ventral hernias]. J Chir (Paris). 2004 Nov;141(6):366-70. doi: 10.1016/s0021-7697(04)95361-6. No abstract available. French. PMID 15738845
- [Background] Proske JM, Vons C. [Laparoscopic treatment of ventral hernias]. J Chir (Paris). 2004 Nov;141(6):360-4. doi: 10.1016/s0021-7697(04)95360-4. French. PMID 15738844